CLINICAL TRIAL: NCT05347004
Title: The Effect of Food on the Pharmacokinetics of a BI 425809 Tablet Formulation Administered as a Single Dose With and Without Food to Healthy Subjects (an Open-label, Randomised, Two-period, Two-sequence Crossover Trial)
Brief Title: A Study in Healthy People to Test How BI 425809 is Taken up in the Body When Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0053; 2021-006659-33 (EudraCT Number)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 425809 fed state (Test, T) then BI 425809 fasting state (Reference, R) (Experimental)
  Interventions: Drug: BI 425809
- BI 425809 fasting state (Reference, R) then BI 425809 fed state (Test, T) (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809 — BI 425809

SUMMARY:
The main objective of this trial is to investigate the potential effect of food on the pharmacokinetics of BI 425809 following administration of the intended Commercial Formulation (iCF) with food (Test treatment, T) and without food (Reference treatment, R).

ELIGIBILITY:
Inclusion criteria:

Subjects will only be included in the trial if they meet the following criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs: Blood pressure (BP), Pulse rate (PR), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subject, or female subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 40 Unites per liter (U/L) and estradiol below 30 nanogram per liter (ng/L) is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 millimetre of mercury (mmHg), or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts

Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 10 Days
Maximum measured concentration of BI 425809 in plasma (Cmax) | Up to 10 Days

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 10 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Madari S, Breithaupt-Groegler K, English BA, Hohl K, Jungnik A, Desch M. Assessing the Effect of Food on the Pharmacokinetics of Iclepertin in Healthy Volunteers: A Phase I, Open-Label, Randomised, Cross-over Trial. Eur J Drug Metab Pharmacokinet. 2025 Sep;50(5):399-408. doi: 10.1007/s13318-025-00956-1. Epub 2025 Jul 17. PMID 40676451
- See also: Related Info — https://www.mystudywindow.com/